CLINICAL TRIAL: NCT02084342
Title: Efficacy and Safety of Desmopressin Combined With Tranexamic Acid on the Blood Loss and Transfusion Need During and After Scoliosis Correction Surgery
Brief Title: Study of DDAVP Combined With TXA on the Blood Loss and Transfusion Need During and After Scoliosis Correction Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Liu Weifeng (Other)
Responsible Party: Sponsor-Investigator, Liu Weifeng, attending doctor, First Affiliated Hospital, Sun Yat-Sen University
Organization: First Affiliated Hospital, Sun Yat-Sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TDS-SYSU-2013
Record Dates: First submitted 2013-12-15; First posted 2014-03-11 (Estimated); Last update posted 2014-03-11 (Estimated); Status verified 2014-03

CONDITIONS: Idiopathic Scoliosis
Keywords: desmopressin; tranexamic acid; blood loss; transfusion need; posterior scoliosis orthopedics
MeSH Terms: conditions — Hemorrhage | interventions — Tranexamic Acid; Sodium Chloride; Saline Solution; Deamino Arginine Vasopressin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group TN (Placebo Comparator): Tranexamic acid and sodium chloride injection at 10mg/kg, IV (in the vein) for 30min, before incision.Then at 1mg/kg/h, IV pump, until the surgery is over.
  Normal saline (NS) 100ml IV for 20min, before incision.
  Interventions: Drug: tranexamic acid and sodium chloride injection; Drug: normal saline
- Group TD (Experimental): Tranexamic acid and sodium chloride injection at 10mg/kg, IV (in the vein) for 30min,before incision.Then at 1mg/kg/h,IV pump,until the surgery is over.
  Desmopressin acetate injection at 0.3μg/kg dissolved in 100ml NS, IV for 20min, before incision.
  Interventions: Drug: tranexamic acid and sodium chloride injection; Drug: desmopressin acetate injection

INTERVENTIONS:
Drug: tranexamic acid and sodium chloride injection — 10mg/kg, IV (in the vein) for 30min, before incision. then at 1mg/kg/h, IV pump, until the surgery is over.
  Other Names: TXA
Drug: normal saline — 100ml, IV for 30min,before incision.
  Other Names: NS
  Arms: Group TN
Drug: desmopressin acetate injection — 0.3μg/kg dissolved in 100ml NS，IV for 30min，before incision.
  Other Names: DDAVP
  Arms: Group TD

SUMMARY:
Intraoperative administration of tranexamic acid (TXA,T) reduces significantly blood loss and blood transfusion requirements during spinal posterior fusion in adolescents with scoliosis. TXA acts mainly by inhibit the plasminogen activator.

Desmopressin (DDAVP ,D) can inhibit the fibrinolytic activity by inducing the release of von Willebrand factor from the endothelial cells. But at the same time, it releases tissue-type plasminogen activator (t-PA), which may cripple its hemostatic effect.

The investigators supposed that if the investigators combine TXA with DDAVP in scoliosis correction surgery, the blood loss and the transfusion need would be reduced significantly.

DETAILED DESCRIPTION:
Intraoperative administration of tranexamic acid (TXA,T) reduces significantly blood loss and blood transfusion requirements during spinal posterior fusion in adolescents with scoliosis. TXA acts mainly by inhibit the plasminogen activator. Desmopressin (DDAVP ,D) can inhibit the fibrinolytic activity by inducing the release of von Willebrand factor from the endothelial cells. But at the same time, it releases tissue-type plasminogen activator (t-PA), which may cripple its hemostatic effect.

The investigators designed a a randomized double-blind clinical combining TXA with DDAVP in scoliosis correction surgery to observe if the blood loss and the transfusion need would be reduced or not.

ELIGIBILITY:
Inclusion Criteria:

* idiopathic scoliosis patients undergoing posterior scoliosis correction surgery
* American society of anesthesiologists(ASA) classification:Ⅰ-Ⅱ
* patients who agreed to participate in this study and has signed the informed consent

Exclusion Criteria:

* blood disease，such as anaemia, idiopathic thrombocytopenic purpura(ITP)
* history of bleeding or ecchymosis
* disorders of laboratory examination on platelets(PLT),prothrombin time(PT),activated partial thromboplastin Time(aPTT),Fibrinogen,D-dimers
* hypertension
* cardiac disease,such as unstable angina, myocardial infarction in recent sis months, cardiac disfunction, congenital heart disease, pulmonary heart disease
* cerebral ischemia
* administering with anticoagulants or nonsteroidal anti-inflammatory drug(NSAID)
* hepatic or renal disease or disfunction
* blood transfusion in recent one month

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-12; Primary Completion 2014-04 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
blood loss | during and 3 days after the surgery
  The blood loss include the volume of blood in suction bottles, the weight of sponges and seroma volume of drainage 3 days after surgery. All fluids added to the surgical field intraoperatively were carefully quantified and deducted from the measured blood loss.

SECONDARY OUTCOMES:
blood transfusion | during and 3 days after the surgery
  The blood transfusion includes all the product needed during and in 3 days after the surgery.

OTHER OUTCOMES:
postoperative complications | up to 24 weeks after the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Wenqi Huang, Ph.D, M.D., Study Chair — First Affiliated Hospital, Sun Yat-Sen University